CLINICAL TRIAL: NCT03078348
Title: Increasing Access to Colorectal Cancer Testing (IACCT) for Blacks
Acronym: IACCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MCC-16501
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma
Keywords: cancer screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Receptor Protein-Tyrosine Kinases; Mass Screening

STUDY DESIGN:
Intervention Model Description: In this modified "block" random assignment, all individuals recruited from the same geographic unit will receive the intervention assigned to that area in order to reduce intervention contamination. Individuals will not be made aware of their randomization (intervention) condition until after baseline assessment. The research assistants will also be assigned at random to work with one geographic area (i.e., one intervention condition) in order to reduce risk of intervention contamination by study staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Psychoeducational Photo Novella (Active Comparator): Fecal Immunochemical Test (FIT) Kit + Culturally targeted Photo Novella Booklet + culturally targeted reminders. This study involves participation at distinct time points:
  1. Baseline
  2. 6 month follow-up
  Interventions: Other: Fecal Immunochemical Test (FIT) Kit; Behavioral: Culturally targeted Photo Novella Booklet
- Standard Brochure Intervention (Active Comparator): FIT Kit + Screen for Life Brochure + standard reminders. This study involves participation at distinct time points:
  1. Baseline
  2. Post 6 month follow-up
  Interventions: Other: Fecal Immunochemical Test (FIT) Kit; Behavioral: Screen for Life Brochure

INTERVENTIONS:
Other: Fecal Immunochemical Test (FIT) Kit — Free FIT Kits distributed at study entry.
Behavioral: Culturally targeted Photo Novella Booklet — Culturally targeted Photo Novella Booklet + culturally targeted reminders. Print materials developed by the Centers for Disease Control and Prevention (CDC)) to provide information about CRC, importance of screening and available screening tests. Timed reminder letters and/or emails intended as a cue to action and as educational boost to facilitate participant screening decision making and screening uptake.
  Arms: Targeted Psychoeducational Photo Novella
Behavioral: Screen for Life Brochure — Screen for Life Brochure + standard reminders. Print materials developed by the Centers for Disease Control and Prevention (CDC)) to provide information about CRC, importance of screening and available screening tests. Timed reminder letters and/or emails intended as a cue to action and as educational boost to facilitate participant screening decision making and screening uptake.
  Arms: Standard Brochure Intervention

SUMMARY:
The purpose of this research study is to compare a new educational material to another widely available educational brochure. The goal is to see if the new educational material will change knowledge and behaviors about colorectal cancer and colorectal screening.

ELIGIBILITY:
Inclusion Criteria:

* Community-based recruitment methods will be used including promotional flyers and word of mouth at locations such as churches, barber shops, civic/community social service centers, senior centers, cultural groups. The flyers will provide brief information and advertise a telephone number for potential participants to call the study office at Moffitt.
* Self identify as Black or African American
* Have no symptoms of colorectal cancer (CRC), or personal diagnosis of CRC or bowel inflammatory disease or related syndromes
* Have not had recent CRC screening per guidelines (never screened or overdue)
* Participants must provide at least two forms of contact information (mailing address, home telephone or cell phone or email address), and contact information of a secondary individual who has a number that is different from the participant (this person may be a relative or friend living with the respondent).
* Spouse or relatives of respondent are potentially eligible.

Exclusion Criteria:

* Individuals who have participated in a colorectal cancer screening (CRCS) research in the past 1 year will not be eligible for this study.
* Additional criteria may apply.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Rate of Fecal Immunochemical Test (FIT) Kit Return Per Study Arm | 6 months post final enrollment
  Fit screening uptake at 6 months. Number of participants who used and returned their FIT Kit, per study arm. A FIT Kit was provided to participants in both study arms for use and return.

SECONDARY OUTCOMES:
Rate of Diagnostic Colonoscopy | Post 6 month follow-up
  Number of participants who participated in a diagnostic colonoscopy, post test kit return.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Gwede, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/